CLINICAL TRIAL: NCT02618720
Title: Intravenous Versus Combined Oral and Intravenous Antimicrobial Prophylaxis for the Prevention of Surgical Site Infection in Elective Colorectal Surgery: A Double-blinded Multicenter Prospective Randomized Controlled Trial
Brief Title: Intravenous Versus Combined Oral and Intravenous Antimicrobial Prophylaxis for the Prevention of Surgical Site Infection in Elective Colorectal Surgery
Acronym: COMBINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0250; 2015-002559-84 (Registry Identifier: 2015-002559-84)
Record Dates: First submitted 2015-11-05; First posted 2015-12-01 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2020-07

CONDITIONS: Elective Colorectal Surgery
Keywords: Antimicrobial prophylaxis; Colorectal surgery; Surgical Site Infection; Postoperative morbidity
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ornidazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ornidazole (Experimental): oral antibiotic prophylaxis using ornidazole, which has a spectrum of activity extended to most anaerobic bacteria and whose pharmacokinetic profile allows a single administration the day before surgery, in addition to intravenous antibiotic prophylaxis could be more effective than intravenous antibiotic prophylaxis alone using cephalosporin in reducing the incidence of SSI after elective colorectal surgery. Given the number of patients operated of colorectal surgery each year, the study is of significant clinical importance
  Interventions: Drug: ornidazole
- placebo (Placebo Comparator): oral antibiotic prophylaxis using ornidazole, which has a spectrum of activity extended to most anaerobic bacteria and whose pharmacokinetic profile allows a single administration the day before surgery, in addition to intravenous antibiotic prophylaxis could be more effective than intravenous antibiotic prophylaxis alone using cephalosporin in reducing the incidence of SSI after elective colorectal surgery. Given the number of patients operated of colorectal surgery each year, the study is of significant clinical importance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ornidazole
  Arms: ornidazole
Drug: Placebo
  Arms: placebo

SUMMARY:
To assess the effects of a combined antimicrobial prophylaxis using oral ornidazole (the day before surgery) and intravenous cephalosporin (before surgical incision) with that of intravenous cephalosporin alone (standard of care) in combination with oral placebo on the incidence of SSI within 30 days after elective colorectal surgery.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is a major cause of nosocomial infection in surgical patients, with the highest rates being reported (ranging from 15% to 30%) in colorectal surgery. SSI is an independent predictor of postoperative mortality and is associated with longer hospital stay, a 5-fold likelihood of postoperative readmission and a 2- to 3-fold increase in costs of care. Given the high prevalence and financial burden associated with SSI, American and European guidelines have been issued providing evidenced-based recommendations for the prevention of postoperative SSI. However, the prevalence of SSI remains high despite adherence to these guidelines and the application of evidence-based preventive measures.

Risk factors for SSI, whether modifiable or not, are mainly related to the patient condition (including age, severe comorbidity, diabetes, nutritional status, steroid use, smoking, and immunosuppression) and/or the surgical procedure (especially the surgical duration and skin disinfection). The prevention of SSI consists of several individual measures, and antibiotic prophylaxis covering aerobic and anaerobic bacteria is highly recommended in patients scheduled to elective colorectal resection, with French and European guidelines recommending the administration of intravenous cephalosporin within 30 minutes before surgical incision.

Recent data from retrospective studies and two meta-analyses of clinical trials provided compelling arguments that oral antibiotic administration before surgery in addition to conventional intravenous prophylaxis may be useful in further reducing by almost 75% the incidence of SSI (relative risk 0.55 [CI95%: 0.41 to 0.74]) after elective colorectal cancer surgery.

However, most of these studies have limitations precluding extrapolation of data into routine care, especially:

1. prolonged duration of intravenous antibiotic administration, which is no longer recommended in elective surgery;
2. the use of antibiotics for oral prophylaxis whose availability is limited;
3. only a few studies focused specifically on colorectal resection;
4. most studies did not include enhanced recovery after surgery (ERAS) programs, which was found to improve outcome following colorectal surgery, and
5. most studies have used mechanical bowel preparation, which is no longer recommended in colonic surgery while the issue still remains open for rectal surgery.

Investigators hypothesized that oral antibiotic prophylaxis using ornidazole, which has a spectrum of activity extended to most anaerobic bacteria and whose pharmacokinetic profile allows a single administration the day before surgery, in addition to intravenous antibiotic prophylaxis could be more effective than intravenous antibiotic prophylaxis alone using cephalosporin in reducing the incidence of SSI after elective colorectal surgery. Given the number of patients operated of colorectal surgery each year, the study is of significant clinical importance

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Laparoscopic or non-laparoscopic elective colorectal surgery

Exclusion Criteria:

* Non elective colorectal surgery (emergent surgery and/or reintervention or revision of a previous colorectal procedure)
* Significant concomitant surgical procedure (e.g., liver resection for metastasis)
* Bacterial infection at the time of surgery or antimicrobial therapy up to 2 weeks before surgery
* Inflammatory bowel disease
* Severe obesity (defined as a BMI >35 kg/m2)
* Known history of hypersensitivity to β-lactams and imidazoles
* Preoperative severe impairment in renal function (creatinine clearance (MDRD) < 30 ml/min)
* Patients with known colonization with multidrug-resistant digestive bacteria, especially multidrug-resistant gram-negative bacteria (requiring specific infection control measures)
* Allergy to lactose, galactose intolerance, Lapp lactase deficiency or glucose/galactose malabsorption (rare metabolic disease)
* Pregnant women, breastfeeding women, women of childbearing age without effective contraceptive- Refusal to participate or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
occurrence of any SSI within 30 days after surgery. | 30 days after surgery
  The primary end point of the trial is the occurrence of any SSI within 30 days after surgery. SSI will be classified as superficial, deep and/or organ-space infection according to validated and well-defined criteria developed by the Centers for Disease Control and Prevention (CDC).

SECONDARY OUTCOMES:
Incidence of individual types of SSI according to the group of treatment | 30 days after surgery
  Incidence of individual types of SSI (superficial incision infection, deep incision infection and organ-space infection) according to the group of treatment, 30 days after surgery
Number of postoperative complications | 30 days after surgery
  Using the Dindo and Clavien classification
Number of surgical complications: anastomotic leakage and the need for abdominal reoperation and/or radiological intervention | 30 days after surgery
Duration of hospital stay | 30 days after surgery
  Including hospital stay of patients who are readmitted after surgery
All-cause mortality | 30 days after surgery
All-cause mortality | 90 days after surgery
Time to introduction of adjuvant chemotherapy related to SSI | 30 days after surgery
Postoperative syndrome of systemic inflammatory response (Infectious complications) | 30 days after surgery
  Number of Postoperative syndrome of systemic inflammatory responses, in each group
Sepsis (Infectious complications) | 30 days after surgery
  Number of Sepsis, in each group
Septic shock (Infectious complications) | 30 days after surgery
  Number of Septic shocks, in each group
Arrhythmia (Cardiovascular complications) | 30 days after surgery
  Number of arrhythmias, in each group
Myocardial infarction (Cardiovascular complications) | 30 days after surgery
  Number of myocardial infarctions, in each group
Acute cardiac failure (Cardiovascular complications) | 30 days after surgery
  Number of acute cardiac failures, in each group
Pneumonia (Respiratory complications) | 30 days after surgery
  Number of pneumonias, in each group
Need for postoperative reventilation (Respiratory complications) | 30 days after surgery
  Number of postoperative reventilations (intubation and/or non-invasive mechanical ventilation), in each group
Renal dysfunction | 30 days after surgery
  Number of Renal dysfunctions in each group. Defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) classification
Time to initiation of adjuvant chemotherapy | 30 days after surgery
  Comparaison of time to initiation of adjuvant chemotherapy between the 2 groups
Need for hospital readmission | 30 days after surgery
  Number of hospital readmissions, in each group
Unexpected admission to intensive care unit | 30 days after surgery
  Number of Unexpected admissions to intensive care unit, in each group
Hospital free days | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942
- [Derived] Futier E, Jaber S, Garot M, Vignaud M, Panis Y, Slim K, Lucet JC, Lebuffe G, Ouattara A, El Amine Y, Couderc P, Dupre A, De Jong A, Lasocki S, Leone M, Pottecher J, Pereira B, Paugam-Burtz C; COMBINE study group. Effect of oral antimicrobial prophylaxis on surgical site infection after elective colorectal surgery: multicentre, randomised, double blind, placebo controlled trial. BMJ. 2022 Nov 3;379:e071476. doi: 10.1136/bmj-2022-071476. PMID 36328372
- [Derived] Vignaud M, Paugam-Burtz C, Garot M, Jaber S, Slim K, Panis Y, Lucet JC, Bourdier J, Morand D, Pereira B, Futier E; COMBINE trial management committee. Comparison of intravenous versus combined oral and intravenous antimicrobial prophylaxis (COMBINE) for the prevention of surgical site infection in elective colorectal surgery: study protocol for a multicentre, double-blind, randomised controlled clinical trial. BMJ Open. 2018 Apr 12;8(4):e020254. doi: 10.1136/bmjopen-2017-020254. PMID 29654027